CLINICAL TRIAL: NCT00852254
Title: Validation of a Novel, Minimally Invasive Ultrasound Indicator Dilution Technique for Measuring Cardiac Index in Critically Ill Children
Brief Title: Validation of Minimally Invasive Ultrasound Indicator Dilution Technique in Critically Ill Children
Status: Completed | Type: Observational
Sponsor: Transonic Systems Inc. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: TSI-C-COSTATUS-6A-H; 2R44HL061994-04A2 (NIH)
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Cardiac Output
Keywords: Cardiac Index; Ultrasound Dilution; Accuracy of ultrasound dilution cardiac index.

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A novel method to measure cardiac index based on ultrasound indicator dilution technology (UIDT) has been developed by Transonic Systems Inc. (Ithaca, NY, USA). The method overcomes many of the limitations that have plagued the existing techniques used to measure cardiac index in critically ill children.

In the proposed investigation, the investigators hope to validate a novel application of an existing technology in critically ill infants and children. The primary aim of this study is to determine the accuracy of cardiac index measured by UIDT when compared to the gold-standard Fick technique. The primary hypothesis is that the average of three consecutive measurements of cardiac index by UIDT will be accurate when compared to the Fick technique. Secondary aims will be to determine the precision of the measurement, the feasibility of the technique with regards to time required and any complications encountered. An exploratory secondary aim of this study is to determine whether central blood volume (CBV) derived from indicator transit time (ITT) correlates with central venous pressure (CVP) and echocardiography derived measures of preload.

ELIGIBILITY:
Inclusion Criteria:

* Age: less than 18 years.
* Admission to the CICU (Cardiac Intensive Care Unit) (8S) or MISICU (Medical-Surgical Intensive Care Unit) (7S) of the Children's Hospital Boston.
* Presence of a central venous catheter with its tip in the superior vena cava or a catheter in the pulmonary artery, documented by radiography.
* Requirement for mechanical ventilation via an endotracheal or tracheostomy tube.
* Presence of an arterial catheter.
* Patients must have a two ventricle circulation.

Exclusion Criteria:

* Endotracheal tube leak of greater than 10%.
* A significant air leak around the endotracheal tube makes VO2 impossible to measure.
* Presence of relevant intracardiac shunt.
* Intracardiac shunt will decrease the area under the arterial dilution curve unpredictably, making cardiac index calculations unreliable.
* A patent foramen ovale and a single ventricular septal defect less than or equal to 2mm or an atrial septal defect less than or equal to 3mm will be considered irrelevant for the purposes of this study.
* Previous enrollment in an incompatible research study.
* Current or prior diagnosis of heparin induced thrombocytopenia.
* A small amount of heparin is required to flush the extracorporeal AV (Arteriovenous) loop that is required for the measurements.
* Pneumothorax with ongoing air leak.
* An air leak will invalidate the measurement of VO2.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients (less than 18 years of age) with in situ arterial and central venous catheters.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2008-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To determine the accuracy of cardiac index measured by ultrasound dilution when compared to the gold-standard Fick technique. | 5-8 minutes minimum

SECONDARY OUTCOMES:
To determine the precision and feasibility of the measurements. Also to determine whether central blood volume (CBV) measured by ultrasound dilution correlates with central venous pressure (CVP) and echocardiography derived preload measures. | 5-8 minutes minimum

CONTACTS AND LOCATIONS:
Overall Officials: Satish Rajagopal, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krivitski NM, Kislukhin VV, Thuramalla NV. Theory and in vitro validation of a new extracorporeal arteriovenous loop approach for hemodynamic assessment in pediatric and neonatal intensive care unit patients. Pediatr Crit Care Med. 2008 Jul;9(4):423-8. doi: 10.1097/01.PCC.0b013e31816c71bc. PMID 18496416